CLINICAL TRIAL: NCT04923477
Title: Mechanisms of Exercise for Rotator Cuff Tendinopathy / Subacromial Pain Syndrome
Brief Title: Therapeutic Exercise for Rotator Cuff Tendinopathy / Subacromial Pain Syndrome - Outcomes and Mechanisms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Lori Michener, Principal Investigator, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-20-00994
Record Dates: First submitted 2021-06-06; First posted 2021-06-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Tendinosis; Rotator Cuff Tendinitis; Rotator Cuff Injuries; Subacromial Pain Syndrome
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: The proposed research will be a prospective longitudinal cohort laboratory experimental design to examine mechanisms of a single bout and 2, 4, and 8 weeks of therapeutic exercise in participants with rotator cuff tendinopathy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Group (Experimental): Therapeutic exercise of resistance and mobility training delivered by a trained health professional x 8 weeks.
  Interventions: Other: Therapeutic Exercise for Rotator Cuff Tendinopathy / Subacromial Pain Syndrome

INTERVENTIONS:
Other: Therapeutic Exercise for Rotator Cuff Tendinopathy / Subacromial Pain Syndrome — Therapeutic exercise of resistance and mobility via a combination of HEP and in-person/virtual visits 5 days/ wk. Exercise program instruction in person, then 2-3 visits /wk x 8 wks (in-person or virtual) with a trained professional for the progression of exercises. Adherence to exercise will be measured daily via text and recorded in a mobile app. Patients will start with Phase 1 exercises of shoulder external & internal rotation, scapular stabilization, and active shoulder elevation; resistance levels of elastic bands will be assigned and progressed based on patient-reported shoulder pain and perceived difficulty. Patients will be advanced to Phase 2 when they complete Phase 1. The exercise protocol will be delivered with the methods previously published by Tate, 2010 and Mintken 2016.

SUMMARY:
Rotator cuff tendinopathy, one of the pathologies identified as part of the cluster of shoulder symptoms known as subacromial pain syndrome, is a common musculoskeletal shoulder condition. Resolution of pain and disability is poor despite treatment, with only about 50% reporting full recovery at 12 - 18 months. Prior studies suggest therapeutic exercise when used alone and with other interventions can have positive outcomes; however, not all patients with rotator cuff tendinopathy respond. Few studies have assessed the effects of exercise for individuals with chronic pain, especially brain driven mechanisms, thought to play a key role. In this study, we will use brain imaging to understand the mechanisms, identify predictors of a positive response to exercise, and the relationship to biomechanical and pain-related factors in patients with RC tendinopathy. The findings from this study will optimize the delivery and treatment response to exercise for individuals with shoulder pain.

DETAILED DESCRIPTION:
Theoretical models propose the development of shoulder pain from an acute injury or repetitive motion seen in sports and certain work environments. Repetitive motions, in combination with altered muscle activity and altered movement strategies, may lead to damage of the rotator cuff structures resulting in local shoulder pain. Emerging evidence supports the hypothesis that localized pain may result in chronic centralized pain over time through central sensitization. Central nervous system changes, specifically those at the level of the brain have been shown to play a role in chronic pain. Neurophysiological mechanisms have been shown to predict symptom progression in other chronic pain conditions. Despite a large body of evidence that therapeutic exercise, mechanisms leading to pain relief are still not well understood. Studies identify a critical role of exercise in modulating excitation and inhibition of key pain centers in the central nervous systems. However, limited evidence exists as to the mechanisms of exercise in the management of patients with chronic pain with therapeutic exercise.

ELIGIBILITY:
Inclusion Criteria:

1. the clinical diagnosis for RC tendinopathy will be made with positive 3 of 5 tests: Hawkins-Kennedy, Neer, painful arc, empty can, external rotation resistance test
2. pain ≥ 3/10 on a numeric pain rating scale
3. age: 18 - 45 years
4. Participant must read, sign and date the appropriate Informed consent document.
5. Participant BMI ≤ 30

Exclusion Criteria:

1. Insufficient ability to comprehend and complete the questionnaires,
2. Inability to attend sessions,
3. Prior surgery of shoulder, neck or thoracic spine,
4. Primary complaint of neck or thoracic pain,
5. Diagnosis of cervical spinal stenosis,
6. Any serious spinal and shoulder pathology: infections, arthrosis, rheumatic disorders, acute fractures, shoulder dislocation, osteoporosis, or tumors,
7. Central Nervous System involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman and/or Babinski reflexes,
8. two or more neurologic signs of nerve root compression to include myotomal weakness, positive muscle stretch reflex, and dermatomal sensory loss,
9. any shoulder or arm pain with cervical spine tests of Spurling's Test, cervical rotation to the ipsilateral side, or axial compression test, or
10. primary adhesive capsulitis defined by passive range of motion loss >50% as compared bilaterally of shoulder external rotation, internal rotation, or elevation.
11. Has a device or other condition that is not safe for MRI, including pacemakers.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pennsylvania Shoulder Score (PENN) | Baseline, 2 weeks, 4 weeks, 8 weeks, 26 weeks and 52 weeks
  The PENN is a self-report measure of pain, satisfaction with shoulder use, and function.
  The pain section has 3 questions of pain at rest, with normal daily activities, and with strenuous activities. The disability section has 20 items rated on a 4-category Likert scale for difficulty (0=cannot do at all, 1=much difficulty, 2=some difficulty, 3=no difficulty, and x=did not do before injury). The satisfaction section is 1 question, rating satisfaction with shoulder use on a 0-10 numeric scale (10 = fully satisfied).

SECONDARY OUTCOMES:
Functional Magnetic Resonance Imaging (fMRI) | Baseline, 2 weeks, 4 weeks, and 8 weeks
  A high resolution structural image will be acquired from each participant with a magnetization-prepared rapid gradient-echo (MP-RAGE) sequence, with a repetition time (TR) = 2200 ms, echo time (TE) = 3.26 ms, slice thickness = 1 mm, 176 slices, 256 × 256 voxel matrices, and 13 mm voxel size. Resting state scans will be acquired while participants rest with eyes closed for 10 min in 40-slice whole brain volumes, with slice thickness = 4 mm, TR = 2000 ms, TE = 28 ms, and flip angle = 77°. Imaging during the rotator cuff muscle activation will be performed by having the participant perform muscle activation tasks for the deltoid and rotator cuff while lying supine in the MRI scanner.
Shoulder Kinematics and Muscle Activity | Baseline, 2 weeks, 4 weeks, and 8 weeks
  Shoulder kinematics of the humerus, thorax, and scapula will be assessed. Muscle activity will be assessed of the rotator cuff (supraspinatus and infraspinatus), deltoid, upper, lower, and middle trapezius, and serratus anterior muscles.
Pain pressure threshold (PPT) | Baseline, 2 weeks, 4 weeks, and 8 weeks
  PPT will be measured using a mechanical pressure algometer (Wagner Instruments, Greenwich, CT) with a flat rubber covered 1 cm2 round force gage over the bilateral deltoids and anterior tibias
OSPRO- Yellow Flags | Baseline, 2 weeks, 4 weeks, 8 weeks, 26 and 52 weeks.
  The Optimal Screening for Prediction of Referral and Outcome (OSPRO) is designed to assess pain-associated psychological distress. The OSPRO-YF includes items from pain vulnerability domains (negative affect and fear-avoidance) and pain resilience domains (positive affect and self-efficacy) to identify pain associated psychological distress. We will use the 17-item version of the OSPRO-YF tool. A summary score can be created by summing all item responses from the original parent questionnaires on the original scale, with pain-resilience items reverse scored, providing a potential score range of 6 to 89, with higher scores indicating higher psychological distress. Scores for each of the 11 original parent questionnaires used to create the OSPRO-YF will also be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Michener, PT, ATC, PhD, Principal Investigator — University of Southern California
Locations (1):
- Clinical Biomechanics Orthopedic and Sports Outcomes Research Laboratory, Los Angeles, California, United States